CLINICAL TRIAL: NCT07028489
Title: Prospective External Control Cohort In Patients With Newly Diagnosed Advanced or Metastatic EGFR Mutant Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: N-Power Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: NPM-002
Record Dates: First submitted 2025-06-09; First posted 2025-06-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: metastatic; advanced
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osimertinib plus chemo, or other regimens: Osimertinib plus chemo, or other regimens in the metastatic setting initiated on or after January 1, 2024
- Osimertinib monotherapy: Osimertinib monotherapy for newly diagnosed mNSCLC

SUMMARY:
The objective of this study is to build a prospective cohort in patients with locally advanced or metastatic NSCLC with common EGFR mutations. In NPM-002, there will be standardized data collection at baseline, on-treatment and at discontinuation of therapy. Patients who enroll prior to initiation of osimertinib treatment (~30%) will undergo imaging with standardized intervals.

ELIGIBILITY:
INCLUSION CRITERIA

* Be ≥18 years of age at the time of informed consent
* Evidence of a confirmed diagnosis of EGFR mutant (EGFR exon 19del or EGFR exon 21 L858R) locally advanced or metastatic NSCLC diagnosed on Jan 1st 2024 or later.

EXCLUSION CRITERIA

* ECOG≥2 at diagnosis of advanced or metastatic NSCLC
* Evidence of prior treatment with osimertinib, amivantamab or lazertinib. For the planned selection and analysis of external controls, further eligibility criteria will be applied according to the COPERNICUS SAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with EGFR mutant locally advanced or metastatic NSCLC diagnosed from Jan 1st 2024 until the enrollment period ends.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Assess real world progression-free survival in patients with locally advanced or metastatic NSCLC treated with first line osimertinib | From the index date (date of initiation of first line treatment for metastatic disease) until date of progression or date of death whichever comes first, assessed up to 100 months)

SECONDARY OUTCOMES:
Assess overall survival in patients with locally advanced or metastatic NSCLC treated with first line osimertinib | From the index date (date of initiation of first line treatment for metastatic disease) until death, as assessed up to 100 months
Assess time to treatment discontinuation in patients with locally advanced or metastatic NSCLC treated with first line osimertinib | From the index date (date of initiation of first line treatment for metastatic disease) until treatment discontinuation, as assessed up to 100 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Pacific Cancer Care, Monterey, California
  - Bayhealth Cancer Center- Kent, Dover, Delaware
  - Bayhealth Cancer Center- Sussex, Milford, Delaware
  - Northwest Oncology & Hematology, Elk Grove Village, Illinois

IPD SHARING:
Plan to Share IPD: Undecided